CLINICAL TRIAL: NCT03236753
Title: Clinical Research on the Efficacy and Safety of Thread-embedding Acupuncture for Treatment of Herniated Intervertebral Disc of Lumbar Spine; A Multicenter, Randomized, Patient-assessor Blinded, Controlled, Parallel Clinical Trial
Brief Title: Clinical Research on the Efficacy of Thread-embedding Acupuncture on Herniated Intervertebral Disc of Lumbar Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); DongGuk University (Other); Daegu Korean Medicine Hospital of Daegu Haany University (Other)
Responsible Party: Principal Investigator, Byung-Kwan Seo, PhD., KMD, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHNMCOH 2016-09-006
Record Dates: First submitted 2017-07-25; First posted 2017-08-02 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Disc Herniation
Keywords: Thread-Embedding Acupuncture; Herniated Intervertebral Disc of Lumbar Spine; Low Back Pain; Radiculopathy
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain; Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thread-Embedding Acupuncture (TEA) (Experimental): The TEA group will be treated once a week for 8 weeks, using 29G x 40mm or 29G x 60mm TEA on predefined 23 acupoints selected by expert group according to STRICTA. All other treatment affecting the outcomes will be prohibited during the trial period. All therapeutic procedure will be performed by acupuncture specialists who have received training for the consensus of multicenter.
  Interventions: Procedure: Thread-embedding Acupuncture (TEA)
- Sham Thread-Embedding Acupuncture (STEA) (Sham Comparator): The STEA group will be treated once a week for 8 weeks, using 29G x 40mm or 29G x 60mm sham TEA on predefined 23 acupoints selected by expert group according to STRICTA.
  Interventions: Procedure: Sham Thread-embedding Acupuncture (STEA)

INTERVENTIONS:
Procedure: Thread-embedding Acupuncture (TEA) — The acupoints and size of TEA are as follows:
  1. Both EX-B2 of herniated intervertebral disc level, its upper level and its lower level (6 acupoints): perpendicular insertion, 4cm
  2. Both BL24: transverse insertion toward L1 level along the erector muscle of spine, 6cm
  3. Both BL25: transverse insertion toward iliac crest, 4cm
  4. Both BL26: transverse insertion toward L1 level along the erector muscle of spine, 6cm
  5. Both BL26: oblique insertion toward iliolumbar ligament, 6cm
  6. Both EX-B7: oblique insertion toward gluteus medius muscle, 6cm
  7. Both BL28: oblique insertion toward sacroiliac ligament, 6cm
  8. Both GB30: perpendicular insertion, 6cm
  9. Symptomatic side GB34, BL57 and ST36: oblique insertion toward foot, 4cm
  Arms: Thread-Embedding Acupuncture (TEA)
Procedure: Sham Thread-embedding Acupuncture (STEA) — All procedure of STEA group, including acupoints and size of TEA will be same as that of TEA group. However, thread-removed TEA will be used for STEA group instead of normal TEA, and removing procedure of thread will be performed aseptic and secretly for patient-blinding and prevention of infection.
  Arms: Sham Thread-Embedding Acupuncture (STEA)

SUMMARY:
This clinical trial is designed to evaluate the efficacy and safety of thread-embedding acupuncture for treatment of lumbar herniated intervertebral disc (L-HIVD) by assessing pain, function, and quality of life.

DETAILED DESCRIPTION:
Seventy patient between the ages of 19 and 70 with L-HIVD will be recruited by eligibility criteria and randomly allocated to the thread-embedding acupuncture (TEA) group and sham thread-embedding acupuncture (STEA) group. Both groups will receive treatment on predefined 23 acupoints once a week for 8 weeks, and needle with thread removed will be used in STEA group instead of normal TEA. 100 mm visual analogue scale (VAS) for low back pain will be assessed as a primary outcome. Also, 100mm VAS for radiating pain, Oswestry disability index (ODI), Rolland Morris disability questionnaire (RMDQ), EQ-5D-5L and global perceived effect (GPE) will be measured as secondary outcomes. All the outcomes will be assessed at baseline, 4 weeks after screening, treatment end (8 weeks, primary end point) and follow-up sessions (12 and 16 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 19-70
2. Radiating pain matched with severer abnormality than bulging shown by CT or MRI on lumbar spine
3. 40 or higher low back pain on 100mm pain VAS
4. Volunteers who agree to participate and sign the Informed Consent Form, following a detailed explanation of clinical trials

Exclusion Criteria:

1. Congenital abnormalities or surgical history on lumbar regions
2. Red flag signs that may be suspected of cauda equina syndrome, such as bladder and bowel dysfunction or saddle anesthesia
3. Tumor, fracture or infection in lumbar regions
4. Injection treatment on lumbar regions within 1 week
5. Psychiatric disorder currently undergoing treatment such as depression or schizophrenia
6. Inappropriate condition for thread-embedding acupuncture due to skin disease or hemostatic disorder (PT INR > 2.0 or taking anticoagulant)
7. Other diseases that could affect or interfere with therapeutic outcomes, including severe gastrointestinal disease, cardiovascular disease, hypertension, diabetes, renal disease, liver disease or thyroid disorder
8. Contraindication of acetaminophen including intercurrent disease, hypersensitivity reaction or other medication
9. Pregnant women or other inappropriate condition for thread-embedding acupuncture
10. Heavy drinking (more than 3 cups per day) that could cause hepatotoxicity with acetaminophen

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline 100mm Pain Visual Analogue Scale (VAS) for low back pain at Week 8 | Week 1 (Baseline), Week 4, Week 8 (Primary end point, Treatment end), Week 12, Week 16 (F/U)
  Measurement instrument for subjective pain

SECONDARY OUTCOMES:
100mm Pain Visual Analogue Scale (VAS) for radiating pain | Week 1 (Baseline), Week 4, Week 8 (Treatment end), Week 12, Week 16 (F/U)
  Measurement instrument for subjective pain
Oswestry Disability Index (ODI) | Week 1 (Baseline), Week 4, Week 8 (Treatment end), Week 12, Week 16 (F/U)
  Validated questionnaire for disability of low back pain.
EuroQol-5 dimensions-5 level (EQ-5D-5L) | Week 1 (Baseline), Week 4, Week 8 (Treatment end), Week 12, Week 16 (F/U)
  Standardized instrument for generic health status
Roland-Morris Disability Questionnaire (RMDQ) | Week 1 (Baseline), Week 4, Week 8 (Treatment end), Week 12, Week 16 (F/U)
  Health status measure for low back pain
Global Perceived Effect (GPE) | Week 4, Week 8 (Treatment end), Week 12, Week 16 (F/U)
  Assessment of change in the patient's chief complaint

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Kwan Seo, PhD., KMD, Principal Investigator — Kyunghee University Medical Center
Locations (4):
- South Korea (4):
  - Dongguk University Bundang Oriental Hospital, Seongnam-si, Gyeonggi-do
  - Daegu Korean Medicine Hospital of Daegu Haany University, Daegu
  - Kyunghee University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goo B, Ryoo DW, Kim EJ, Nam D, Lee HJ, Kim JS, Park YC, Baek YH, Seo BK. Clinical research on the efficacy and safety of thread-embedding acupuncture for treatment of herniated intervertebral disc of the lumbar spine: a protocol for a multicenter, randomized, patient-assessor blinded, controlled, parallel, clinical trial. Trials. 2018 Sep 10;19(1):484. doi: 10.1186/s13063-018-2864-4. PMID 30201029